CLINICAL TRIAL: NCT03691675
Title: Prospective Clinical Research on Safety and Efficacy of Drug Coated Balloon in de Novo Coronary Lesion With Diameters Larger Than 2.75 mm Under OCT Guidance
Brief Title: DCB in de Novo Coronary Lesion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Liu Bin, Chief of Department, Second Hospital of Jilin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SecondJilinU-3
Record Dates: First submitted 2018-09-28; First posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Drug-coated Balloon
Keywords: Drug-coated balloon; restenosis; dissection

STUDY DESIGN:
Intervention Model Description: Patients with de novo lesion whose radiography showed that target lesion diameter stenosis is ≥50%, reference diameter is ≥2.75mm and who agreed with the Drug coated balloon dilatation therapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drug coated balloon (Experimental): Patients with de novo lesion whose radiography showed that target lesion diameter stenosis is ≥50%, reference diameter is ≥2.75mm and who agreed with the Drug coated balloon dilatation therapy
  Interventions: Device: Drug coated balloon

INTERVENTIONS:
Device: Drug coated balloon — Patients with de novo lesion whose radiography showed that target lesion diameter stenosis is ≥50%, reference diameter is ≥2.75mm and who agreed with the Drug coated balloon dilatation therapy

SUMMARY:
Intro-stent restenosis, bifurcation lesions and small vascular lesion with diameter <2.75mm is the indication of drug coated balloon. In the era of traditional coronary artery balloon dilatation, it is believed that muscle fiber of coronary artery great vessels is more abundant than that of small vessels, and elastic recoil and dissection are easier to appear upon dilatation, which will result in acute vascular occlusion and restenosis, so it is not recommended for great vessels to only receive PTCA therapy. But for patients with good angiography result without combination of serious dissections after predilation, the acute thrombosis seems to be a key factor for acute vascular occlusion. Traditional antiplatelet drug doesn't have a good effect, but the application of new-generation antiplatelet drug (clopidogrel, ticagrelor and tirofiban) has greatly reduced the occurrence rate of acute thrombosis. Therefore, under the guarantee of fully antiplatelet action of new-generation antiplatelet drug, for the patients with good angiography result without combination of serious dissections after predilation, Drug coated balloon seems to be an alternative of the stent. This research is to verify the safety and efficacy of Drug coated balloon in de novo coronary artery lesion with vascular diameter ≥2.75mm.

DETAILED DESCRIPTION:
Stable or unstable angina patients who accept drug coated balloon dilatation therapy with diameter stenosis≥50%, reference diameter≥2.75mm will be enrolled. OCT examination should be carried out after radiography, predilation, Drug coated balloon dilatation and follow-up.

For target lesion, balloon should be used for predilation (the ratio of balloon diameter to vascular diameter being 0.8-1.0:1), and for good predilation effects, high pressure balloon, cutting balloon, dual-wire balloon and spines balloon can be adopted. OCT examination should be carry out after balloon satisfactory predilation. Satisfactory predilation radiography result is residual stenosis≤30%,TIMI 3 flow without major dissections (type C or higher) in NHLBI classification. OCT satisfactory result is residual stenosis≤30% without dissection, or with dissection but the dissection angle is ≤90°. Then carry out DCB balloon dilatation therapy. The ratio of balloon diameter to vascular diameter is 0.8-1.0:1, and both ends of DCB exceed the preprocessing area of lesion for 2-3mm, thus avoiding the occurrence of geographical mismatch. Dilation pressure is 8-10atm, lasting for at least 30s. Each DCB catheter can be used once only.

ELIGIBILITY:
Inclusion Criteria

* At the age of 18-80 (18 and 80 included)
* The female at reproductive age shouldn't get pregnant or plan to get pregnant during the research
* Patients must agree to accept 3-month angiography follow-up
* Patients must agree to accept clinical follow-up on 30-day, 60-day and 90-day after operation
* Psychologically and linguistically, patients could have an understanding of the research purpose, revealing sufficient compliance with the research proposal. The patients' provision of the informed consent represents that the patient accepts the risks and benefits described in the informed consent.
* Target lesion diameter stenosis is ≥50%, and reference vascular diameter is ≥2.75mm
* De novo coronary lesion
* Type A lesion

Exclusion criteria

* Patients with myocardial infarction within one week
* Patients with congestive heart failure or severe NYHAIV heart failure
* Patients with severe valvular heart disease
* The female in pregnancy or lactation period
* Patients whose life expectancy don't exceed 1 year or who might have difficulty in clinical follow-up
* Patients who are of bleeding physique or forbidden to administer anticoagulants or antiplatelet drugs
* Patients who suffered from cerebral stroke within 6 months prior to surgery
* Patients who are involved in any other clinical trials
* Patients who fail to satisfy angiography conditions due to currently suffering from or previously undergoing severe renal failure (GFR<30ml/min)
* Patients who underwent heart transplantation
* Patients who are deemed inappropriate for inclusion by the researcher due to other reasons
* Lesion of left main coronary artery
* Double vessel or triple vessel disease needed to be interventional treated
* Double vessel or triple vessel disease needed to be interventional treated
* Patients who are intolerant of aspirin and/or clopidogrel, have the medical history of neutrocytopenia or thrombocytopenia, or are forbidden to administer clopidogrel due to severe hepatic insufficiency
* Patients with known hypersensitivity
* Patients with the history of leukopenia (white blood cell count<3x109/L for over 3 days), or neutrocytopenia (ANCs <1,000 neutrophils/mm3 for over 3 days) or thrombocytopenia (blood platelets<100,000/mm3)
* Patients having the history of peptic ulcer or gastrointestinal bleeding within the past 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Lumen loss in advanced stage of lesion segments within 3 months | 3 months
  Lumen loss in advanced stage of lesion segments within 3 months

SECONDARY OUTCOMES:
Success rate of interventional therapy (including device success rate, lesion success rate and clinical success rate) | 3 months
Occurrence rate of dissection after procedure | 3 months
Binary restenosis rate 3 months after procedure | 3 months
Cardiovascular clinical composite endpoints related to device at the time of 30 days, 60 days and 90days after the surgery include cardiac death, target vessel myocardial infarction and target lesion revascularization driven by clinical symptoms, | 3 months
Cardiovascular clinical composite endpoints related to patients at the time of 30 days, 60 days and 90 days after the surgery include all-cause mortality, all myocardial infarction and any revascularization | 3 months
ARC-defined occurrence rate of thrombotic events (identified, probable and non-excluded thrombosis during acute, subacute and advanced stage) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Bin Liu, Doctor, Principal Investigator — Second Hospital of Jilin University